CLINICAL TRIAL: NCT07052175
Title: Prevention of Relapse in Behavioral Disorders: Study Protocol of a Randomized Control Trial
Brief Title: Prevention of Relapse in Behavioral Disorders
Acronym: PreCare
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clínica Nuestra Señora de la Paz (Other)
Collaborators: Universidad Carlos III de Madrid (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CPP2022-00953
Record Dates: First submitted 2025-06-18; First posted 2025-07-04 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Substance-related Disorders
Keywords: Substance use disorders; relapse prevention; multidisciplinary treatment; digital health; monitoring
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial, efficacy study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Treatment Group (Active Comparator): Participants in this group will receive the standard multidisciplinary treatment for substance use disorders, including clinical evaluation, medical detoxification, psychological and psychiatric therapy, occupational rehabilitation, and social reintegration, without the use of the digital tool
  Interventions: Behavioral: Standard Multidisciplinary Treatment
- Digital-Assisted Treatment Group (Experimental): Participants in this group will receive the same standard multidisciplinary treatment as Arm 1, complemented by a digital tool designed for real-time monitoring, early relapse detection, and personalized feedback throughout the follow-up phase
  Interventions: Behavioral: Standard Multidisciplinary Treatment; Behavioral: Digital Monitoring Tool

INTERVENTIONS:
Behavioral: Standard Multidisciplinary Treatment — Comprehensive intervention including structured phases: initial assessment, detoxification, withdrawal management, psychological and psychiatric therapy, rehabilitation, and follow-up care. Delivered by a multidisciplinary team according to established clinical protocols.
Behavioral: Digital Monitoring Tool — In addition to standard care, participants will use a mobile application that monitors clinical indicators, detects early signs of relapse risk, and provides personalized alerts and intervention prompts. The tool is designed to support both patients and clinicians in decision-making and therapeutic follow-up.
  Arms: Digital-Assisted Treatment Group

SUMMARY:
This study aims to validate the effectiveness of a digital tool for monitoring and early relapse detection in addiction treatment. It compares outcomes between a traditional multidisciplinary model and the same model enhanced by the technology. The research seeks to demonstrate the tool's added clinical value in improving long-term recovery outcomes.

DETAILED DESCRIPTION:
The primary objective of this research project is to scientifically validate the effectiveness of a technological tool for monitoring and early detection of relapse in addiction treatment. The study will focus on comparing two approaches: the traditional comprehensive multidisciplinary treatment model and the same model enhanced by the integration of a digital technology.

The comprehensive model addresses the biological, psychological, and social dimensions of substance use disorders through a structured sequence of phases: initial assessment, detoxification, withdrawal management, rehabilitation, social reintegration, and follow-up care. The core innovation of this study lies in the implementation of a digital application specifically designed to monitor patients' clinical status, detect early warning signs of relapse, and deliver timely, personalized interventions.

A longitudinal quasi-experimental study will be conducted with a sample of 150 individuals diagnosed with substance use disorders (including alcohol, cocaine, and other stimulants). Validated assessment instruments will be used to evaluate clinical progress, comparing outcomes between patients receiving standard treatment and those receiving the same treatment augmented by the digital tool.

Key outcome variables include reduction in withdrawal symptoms, decrease in craving, improvement in emotional well-being and psychosocial functioning, relapse rates, and patient satisfaction. In addition, the feasibility, acceptability, and clinical utility of the technological tool in therapeutic follow-up will be assessed.

The study is expected to provide empirical evidence on the added value of the digital tool in addiction treatment, with the aim of optimizing existing clinical protocols and enhancing the long-term effectiveness of intervention strategies.

ELIGIBILITY:
Inclusion Criteria:

* Understand spoken and written Spanish.
* Signing the informed consent.
* Own a smartphone with internet access and an iOS or Android operating system.

Exclusion Criteria:

* Institutionalized or incarcerated patients, or those anticipating imminent incarceration, without regular access to mobile phone use.
* Refusal to install the mobile application.
* Inability to understand and sign the informed consent form for any reason.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Biological Verification of Substance Use Relapse via Toxicological Testing: Urinalysis | Throughout the intervention and follow-up phases (baseline to 12 months)
  To objectively identify episodes of relapse (e.g., alcohol or other substance use) during treatment, periodic toxicological screenings will be performed as part of the therapeutic monitoring process. These screenings are conducted by clinical personnel and include urinalysis: detection of recent use of psychoactive substances through urine samples, providing an objective measure of treatment adherence.
Biological Verification of Substance Use Relapse via Toxicological Testing: Breath Alcohol Testing | Throughout the intervention and follow-up phases (baseline to 12 months)
  To objectively identify episodes of alcohol relapse during treatment, periodic toxicological screenings will be conducted as part of the therapeutic monitoring process. These screenings will be carried out by clinical staff and will include Breath Alcohol Testing: measurement of breath alcohol concentration using spirometry-based devices to detect recent alcohol consumption.

SECONDARY OUTCOMES:
WHOQOL-BREF | Baseline, post-treatment (3 months), and follow-up (6 and 12 months)
  A 26-item instrument assessing perceived quality of life across four domains: physical health, psychological well-being, social relationships, and environmental context. Items are rated on a 5-point Likert scale, and domain scores are transformed to a 0-100 scale. Demonstrates good internal consistency, with Cronbach's alpha ranging from 0.69 (physical) to 0.90 (spirituality/religion/personal beliefs).
Purpose in Life Test - Short Form (PIL-10) | Baseline, post-treatment (3 months), and follow-up (6 and 12 months)
  A 10-item self-report scale assessing life purpose and personal meaning, adapted from the original PIL (Crumbaugh & Maholick, 1969). Responses are rated on a 7-point Likert scale, with total scores ranging from 10 to 70. Higher scores reflect greater perceived purpose. The scale includes two dimensions: (a) life satisfaction and meaning, and (b) goals and direction. Shows good psychometric properties (α = .85 overall; .84 for life satisfaction and .69 for goals and purpose).
Patient Health Questionnaire-9 (PHQ-9) | Baseline, post-treatment (3 months), and follow-up (6 and 12 months)
  A 9-item self-report tool assessing depressive symptom severity over the past two weeks, based on DSM-IV criteria. Each item is scored from 0 (not at all) to 3 (nearly every day), yielding a total score of 0-27. A cut-off score of 10 yields sensitivity of 0.78 and specificity of 0.87. Spanish versions show excellent reliability (α = 0.78-0.90), with current data showing α = .93.
Beliefs About Substance Use and Craving Beliefs Questionnaire | Baseline, post-treatment (3 months), and follow-up (6 and 12 months)
  25 items self-report questionnaire designed to assess maladaptive beliefs related to substance use and beliefs about substance craving. Each item is rated on a 5-point Likert scale ranging from "totally disagree" to "totally agree". Higher total scores reflect stronger dysfunctional beliefs associated with substance use (e.g., perceived benefits or inevitability of use). The instrument shows excellent internal consistency (Cronbach's alpha = 0.87).

OTHER OUTCOMES:
Patient Satisfaction with the Digital Application | Post-treatment (3 months)
  27-item ad hoc questionnaire using a 5-point Likert scale (scale from 1 to 5, with 1 being "Not at all" and 5 being "Very much") to assess patient satisfaction with the application's usability, safety, and overall experience. Higher scores indicate greater satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Jesús Muñoz García, PhD, Principal Investigator — Centro San Juan de Dios de Ciempozuelos; Antonio Artés, PhD, Principal Investigator — Department of Signal Theory at Universidad Carlos III; Apolo Zepeda Avilés, Medical Director, Principal Investigator — Hospital San Juan de Dios de Gipuzkoa; Enrique Bermúdez Navas, Psychiatrist, Principal Investigator — Centro Asistencial San Juan de Dios Palencia; Placidia Franco Suárez-Bárcena, Technical Director, Principal Investigator — Centro Asistencial San Juan de Dios Palencia; Rafael Salom Borrás, PhD, Principal Investigator — Clínica Nuestra Señora de la Paz, Orden Hospitalaria San Juan de Dios, Madrid, Spain; Álvaro Pico Rada, Medical Director, Principal Investigator — Clínica Nuestra Señora de la Paz, Orden Hospitalaria San Juan de Dios, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
IPD information will not be shared due to the sensitivity of the data it contains, which could allow for the direct or indirect identification of patients.

REFERENCES:
- [Result] Salom R, Pico Rada A, Munoz Garcia JJ, Garcia-Mieres H, Artes-Rodriguez A. Digital relapse prevention plan for substance use disorders: study protocol for a multicentre randomised controlled trial. BMJ Health Care Inform. 2025 Nov 24;32(1):e101808. doi: 10.1136/bmjhci-2025-101808. PMID 41290251